CLINICAL TRIAL: NCT02573467
Title: Extension of the CBYM338B2203 Phase IIb/III Study to Evaluate the Long-term Efficacy, Safety and Tolerability of Intravenous BYM338 in Patients With Sporadic Inclusion Body Myositis
Brief Title: An Extension Study of the Efficacy, Safety and Tolerability of BYM338 (Bimagrumab) in Patients With Sporadic Inclusion Body Myositis Who Previously Participated in the Core Study CBYM338B2203
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBYM338B2203E1; 2015-001411-12 (EudraCT Number)
Record Dates: First submitted 2015-07-09; First posted 2015-10-09 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-02

CONDITIONS: Sporadic Inclusion Body Myositis
Keywords: sporadic inclusion body myositis,; muscle wasting,; extension study,; BYM338,; bimagrumab,
MeSH Terms: conditions — Myositis, Inclusion Body; Muscular Atrophy | interventions — bimagrumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BYM338/bimagrumab 10 mg/kg (Experimental): Participants received BYM338 10 mg/kg administered via intravenous infusion every 4 weeks for up to a maximum of 8 months after which they entered a 6-month, treatment-free follow-up period.
  Interventions: Drug: Bimagrumab
- BYM338/bimagrumab 3 mg/kg (Experimental): Participants received BYM338 3 mg/kg administered via intravenous infusion every 4 weeks for up to a maximum of 8 months after which they entered a 6-month, treatment-free follow-up period.
  Interventions: Drug: Bimagrumab
- BYM338/bimagrumab 1 mg/kg (Experimental): Participants received BYM338 1 mg/kg administered via intravenous infusion every 4 weeks for up to a maximum of 8 months after which they entered a 6-month, treatment-free follow-up period.
  Interventions: Drug: Bimagrumab
- Placebo (Placebo Comparator): Participants received placebo administered via intravenous infusion every 4 weeks for up to a maximum of 8 months after which they entered a 6-month, treatment-free follow-up period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bimagrumab — BYM338, a 150 mg/mL concentrate for solution for i.v. infusion, was provided in colorless glass vials with a rubber stopper and aluminum flip-off caps.
  Other Names: BYM338
  Arms: BYM338/bimagrumab 1 mg/kg; BYM338/bimagrumab 10 mg/kg; BYM338/bimagrumab 3 mg/kg
Drug: Placebo — Matching placebo to BYM338 was provided in colorless glass vials with a rubber stopper and aluminum flip-off caps.
  Arms: Placebo

SUMMARY:
This extension study will provide data to further evaluate the efficacy, safety, and tolerability of three doses of BYM338 and to assess the long-term effects of BYM338 in patients with sporadic inclusion body myositis. The extension study was planned to consist of a Screening epoch (to assess patient eligibility), followed by a Treatment Period 1 epoch (double-blind and placebo-controlled), and a Treatment Period 2 epoch (open-label). A Post-treatment Follow-up (FUP) epoch was also planned for patients who discontinued prematurely. Patients who complete the core study and qualify for this extension study entered Treatment Period 1 and continued on the study drug to which they were randomized in the core study (either to one of the three bimagrumab doses (1 mg/kg, 3 mg/kg, and 10mg/kg) or placebo) during Treatment Period 1. Thus, Treatment Period 1 was double-blind and placebo-controlled. Participants were to continue in Treatment Period 1 until the dose with the best benefit-risk profile was determined from the core study data and selected (duration of Treatment Period 1 was estimated to be between 6 and 8 months). Once the dose with the best benefit-risk profile was selected, all participants (including those who were receiving placebo) were planned to enter Treatment Period 2 and switch to open-label treatment with bimagrumab at the selected dose. The core study has been completed but since the core study did not meet the primary end point (no bimagrumab dose was identified based on the core study efficacy results) the extension study was terminated as per protocol/sponsor's decision; therefore, no patients had entered Treatment Period 2. Instead, all patients were to return for the End of Treatment Period 1 (EOT1) visit at their next scheduled visit. As per protocol, all patients who discontinued study medication during Treatment Period 1 for any reason, including due to the study having been stopped as per protocol/sponsor's decision, were to have entered and complete the 6-month FUP after their EOT1 visit.

Due to the nature of the design of the core and extension studies and termination of study medication in the extension study, the treatment duration for individual patients varied considerably. Consequently, the number of patients contributing data to the efficacy analyses at Week 104 and later timepoints was decreased.

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed the core study
* Written informed consent must be obtained before any extension study assessment is performed.
* Able to communicate well with the investigator.
* Willing to participate for the entire duration of the extension study with commitment to follow study requirements and procedures.

Exclusion Criteria:

* Women who are pregnant
* Women of child-bearing potential unless they are using highly effective methods of contraception during dosing and for 6 months after the last BYM338 dose.
* Current use of prohibited treatments
* History of severe hypersensitivity reaction in the core study
* History of adverse event(s) (including those from the core study) prior to the start of study drug in the extension study that, in the judgment of the investigator, taking into account the subject's overall status, prevent the subject from entering the extension study
* Clinically significant abnormal liver function tests
* Any medical condition or laboratory finding which, in the opinion of the investigator may interfere with participation in the study, might confound the results of the study, or pose an additional safety risk in administering BYM338

Min Age: 36 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2016-08-17 (Actual); Study Completion 2017-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (37):
- United States (11):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Orange, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Kansas City, Kansas
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
- Australia (3):
  - Novartis Investigative Site, St Leonards, New South Wales
  - Novartis Investigative Site, Cauldfield, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
- Belgium (3):
  - Novartis Investigative Site, Edegem, Antwerpen
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
- Novartis Investigative Site, Copenhagen, Denmark
- Novartis Investigative Site, Paris, France
- Italy (5):
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Rome, Lazio
  - Novartis Investigative Site, Messina, ME
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Padua, PD
- Japan (7):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kumamoto, Kumamoto
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Kodaira, Tokyo
  - Novartis Investigative Site, Wakayama, Wakayama
  - Novartis Investigative Site, Tokushima
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Leiden
- Novartis Investigative Site, Zurich, Switzerland
- United Kingdom (3):
  - Novartis Investigative Site, Salford, Manchester
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newcastle upon Tyne

REFERENCES:
- [Derived] Amato AA, Hanna MG, Machado PM, Badrising UA, Chinoy H, Benveniste O, Karanam AK, Wu M, Tanko LB, Schubert-Tennigkeit AA, Papanicolaou DA, Lloyd TE, Needham M, Liang C, Reardon KA, de Visser M, Ascherman DP, Barohn RJ, Dimachkie MM, Miller JAL, Kissel JT, Oskarsson B, Joyce NC, Van den Bergh P, Baets J, De Bleecker JL, Karam C, David WS, Mirabella M, Nations SP, Jung HH, Pegoraro E, Maggi L, Rodolico C, Filosto M, Shaibani AI, Sivakumar K, Goyal NA, Mori-Yoshimura M, Yamashita S, Suzuki N, Aoki M, Katsuno M, Morihata H, Murata K, Nodera H, Nishino I, Romano CD, Williams VSL, Vissing J, Zhang Auberson L; RESILIENT Study Extension Group. Efficacy and Safety of Bimagrumab in Sporadic Inclusion Body Myositis: Long-term Extension of RESILIENT. Neurology. 2021 Mar 23;96(12):e1595-e1607. doi: 10.1212/WNL.0000000000011626. Epub 2021 Feb 17. PMID 33597289

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants entered extension study treatment period after completing the core study and continued on the study drug to which they were randomized in the core study (one of 3 bimagrumab doses (1mg/kg, 3mg/kg or 10mg/kg) or placebo). Participants discontinued from the treatment period were to enter a 6-month, treatment-free Follow-up Period (FUP).
Pre-assignment Details: All participants (N=211) were discontinued from the double-blind treatment period, 178 of whom entered the FUP. Overall 154 participants completed the FUP and 20 discontinued due to subject/guardian decision and 1 for technical reasons. Three discontinued FUP due to death (one each in the 10mg/kg, 3mg/kg, and placebo groups).
Groups:
- Placebo: Participants received BYM338 1 mg/kg administered via intravenous infusion every 4 weeks for up to a maximum of 8 months after which they entered a 6-month, treatment-free follow-up period.
Period: Double-blind Treatment Epoch
Arm/Group | BYM338/Bimagrumab 10 mg/kg | BYM338/Bimagrumab 3 mg/kg | BYM338/Bimagrumab 1 mg/kg | Placebo
Started (Mean duration of exposure during the extension double-blind treatment period was 197.2 to 212.3 days) | 53 | 52 | 51 | 55
Full Analysis Set | 53 | 52 | 51 | 55
Completed | 0 | 0 | 0 | 0
Not Completed | 53 | 52 | 51 | 55
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 0
Not completed — Study Terminated by sponsor | 50 | 51 | 48 | 55
Period: Post-treatment Follow up Epoch
Arm/Group | BYM338/Bimagrumab 10 mg/kg | BYM338/Bimagrumab 3 mg/kg | BYM338/Bimagrumab 1 mg/kg | Placebo
Started | 41 | 46 | 44 | 47
Completed | 35 | 41 | 34 | 44
Not Completed | 6 | 5 | 10 | 3
Not completed — Death | 1 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 5 | 4 | 9 | 2
Not completed — Technical problems | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BYM338/Bimagrumab 10 mg/kg | BYM338/Bimagrumab 3 mg/kg | BYM338/Bimagrumab 1 mg/kg | Placebo | Total
Number analyzed (Participants) | 53 | 52 | 51 | 55 | 211
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.2 (8.19) | 67.3 (9.04) | 70.0 (7.69) | 69.9 (7.95) | 69.1 (8.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 17 | 19 | 73
  Male | 35 | 33 | 34 | 36 | 138

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and Deaths.
Description: Safety monitoring was conducted throughout the study. AEs starting on or after the day of first administration of extension study drug until last administration of study drug + 56 days are considered. SAEs starting on or after the day of first administration of extension study drug are considered. Deaths which occurred on or after the day of first administration of extension study drug are considered.
Time Frame: to end of study (up to 14 months, including the 6-month treatment-free follow-up period)
Population: Safety set: The safety set consisted of all participants who received at least one dose of study drug during the extension study.
Measure: Number; unit: Participants
Arm/Group | BYM338/Bimagrumab 10 mg/kg | BYM338/Bimagrumab 3 mg/kg | BYM338/Bimagrumab 1 mg/kg | Placebo
Number analyzed (Participants) | 53 | 52 | 51 | 55
Participants
  Adverse events | 48 | 50 | 44 | 49
  Serious adverse events | 12 | 10 | 7 | 8
  Deaths | 1 | 1 | 1 | 2

2. Primary Outcome: Change From Core Study Baseline in 6 Minute Walking Distance Test (6MWD)
Description: The 6MWD test measures the distance (in meters) that a participant can walk in a 6 minute time frame. A positive change from baseline indicates improvement. The efficacy analysis and time points were based on windowed visits relative to the first dose of the double-blind treatment in the core study.
Time Frame: Core study baseline, weeks 52, 78, 104, and >=117
Population: The full analysis set, which consisted of all participants who were assigned to treatment in the core study and who received at least one dose of study drug during the extension, was considered for the analysis. Participants with both core baseline (BL) and post core-BL values for each time point were analyzed for that time point.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | BYM338/Bimagrumab 10 mg/kg | BYM338/Bimagrumab 3 mg/kg | BYM338/Bimagrumab 1 mg/kg | Placebo
Number analyzed (Participants) | 53 | 52 | 51 | 55
meters
  Week 52 (n=53,52,51,54): number analyzed (Participants) | 53 | 52 | 51 | 54
  Week 52 (n=53,52,51,54) | 6.88 (68.948) | 9.48 (81.676) | -14.26 (81.029) | -5.98 (78.817)
  Week 78: number analyzed (Participants) | 52 | 52 | 50 | 54
  Week 78 | -5.25 (122.002) | -9.73 (68.302) | -18.66 (81.536) | -32.78 (96.494)
  Week 104: number analyzed (Participants) | 32 | 34 | 37 | 39
  Week 104 | -22.68 (102.549) | -50.58 (118.012) | -25.08 (95.737) | -61.30 (107.399)
  >=Week 117: number analyzed (Participants) | 2 | 1 | 4 | 1
  >=Week 117 | -206.65 (281.923) | -5.0 (NA) — Standard deviation (SD) does not apply when n = 1. | -53.65 (114.322) | 31.60 (NA) — SD does not apply when n = 1.

3. Secondary Outcome: Change From Core Study Baseline in Quadriceps Quantitative Muscle Testing (QMT) on the Right Side
Description: Quantitative Muscle Testing (QMT) was used to describe the long-term evolution of quadriceps muscle strength on the right side. The QMT was performed using the same portable fixed dynamometry (PFD) used in the core study. A negative change from baseline indicates deterioration. The efficacy analysis and time points were based on windowed visits relative to the first dose of the double-blind treatment in the core study.
Time Frame: Core study baseline, week 52, week 78, week 104 and >=week 117
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: newtons
Arm/Group | BYM338/Bimagrumab 10 mg/kg | BYM338/Bimagrumab 3 mg/kg | BYM338/Bimagrumab 1 mg/kg | Placebo
Number analyzed (Participants) | 53 | 52 | 51 | 55
newtons
  Week 52: number analyzed (Participants) | 48 | 49 | 51 | 55
  Week 52 | -6.29 (31.121) | -19.70 (77.820) | -5.62 (32.245) | -14.22 (27.577)
  Week 78: number analyzed (Participants) | 46 | 49 | 49 | 53
  Week 78 | -9.43 (41.285) | -23.76 (73.729) | -17.04 (25.696) | -21.02 (31.391)
  Week 104: number analyzed (Participants) | 33 | 33 | 37 | 37
  Week 104 | -11.92 (35.243) | -16.99 (34.379) | -18.63 (37.968) | -21.91 (39.985)
  >=Week 117: number analyzed (Participants) | 1 | 1 | 4 | 1
  >=Week 117 | 67.64 (NA) — SD does not apply when n = 1. | 33.38 (NA) — SD does not apply when n = 1. | -19.36 (18.475) | -18.24 (NA) — SD does not apply when n = 1.

4. Secondary Outcome: Change From Core Study Baseline in Sporadic Inclusion Body Myositis (sIBM) Functional Assessment (sIFA) Score
Description: Self-reported physical function was assessed by a newly developed patient reported outcome named sporadic inclusion body myositis (sIBM) functional assessment (sIFA). The sIFA consists of 11 items scored on an 11 point numerical rating scale from 0 (no difficulty) to 10 (unable to do) across 3 domains: upper body functioning, lower body functioning and general functioning. Participants completed the assessment where the recall period was the past week prior to completing the patient reported outcome (PRO). The total score on the sIFA scale ranges from 0 (minimum) to 110 (maximum). Higher values represent a worse outcome. A positive change from baseline indicates deterioration. The efficacy analysis and time points were based on windowed visits relative to the first dose of the double-blind treatment in the core study.
Time Frame: Core study baseline, week 52, week 78, week 104, and >=week 117
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BYM338/Bimagrumab 10 mg/kg | BYM338/Bimagrumab 3 mg/kg | BYM338/Bimagrumab 1 mg/kg | Placebo
Number analyzed (Participants) | 53 | 52 | 51 | 55
score on a scale
  Week 52: number analyzed (Participants) | 53 | 52 | 49 | 52
  Week 52 | -1.34 (15.249) | 1.80 (11.910) | 3.17 (11.380) | 5.16 (13.889)
  Week 78: number analyzed (Participants) | 53 | 51 | 48 | 54
  Week 78 | -0.27 (13.745) | 5.33 (13.099) | 6.52 (12.918) | 7.41 (14.410)
  Week 104: number analyzed (Participants) | 38 | 37 | 35 | 40
  Week 104 | 3.54 (14.998) | 8.04 (16.861) | 5.97 (12.849) | 7.39 (15.580)
  >=Week 117: number analyzed (Participants) | 2 | 1 | 4 | 1
  >=Week 117 | -16.37 (21.857) | 10.91 (NA) — SD does not apply when n = 1. | 1.37 (17.655) | 6.36 (NA) — SD does not apply when n = 1.

5. Secondary Outcome: Estimated Annual Number of Falls Per Participant Within Treatment Group
Description: Participants documented any fall occurrences in a paper diary during the study.
Time Frame: Core baseline to end of extension double-blind treatment (up to a maximum of 32 months)
Population: Safety set: The safety set consisted of all participants who were assigned to treatment in the core study and who received at least one dose of study drug during the extension.
Measure: Number; unit: Annual number of falls per participant
Arm/Group | BYM338/Bimagrumab 10 mg/kg | BYM338/Bimagrumab 3 mg/kg | BYM338/Bimagrumab 1 mg/kg | Placebo
Number analyzed (Participants) | 53 | 52 | 51 | 55
Annual number of falls per participant | 4.164 | 3.879 | 3.480 | 3.835

6. Secondary Outcome: Change From Core Study Baseline in Short Physical Performance Battery (SPPB) Score
Description: The SPPB evaluated lower extremities function by testing gait speed, ability to keep standing balance and time to rise from a chair five times. The sub-score for each test ranged from 0 to 4. The summary score, which was a summation of scores from the 3 tests, ranged from 0 to 12. An increase in score indicates improvement in physical performance. A negative change from baseline indicates deterioration. The efficacy analysis and time points were based on windowed visits relative to the first dose of the double-blind treatment in the core study.
Time Frame: Core study baseline, week 52, week 78, week 104 and >=week 117
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BYM338/Bimagrumab 10 mg/kg | BYM338/Bimagrumab 3 mg/kg | BYM338/Bimagrumab 1 mg/kg | Placebo
Number analyzed (Participants) | 53 | 52 | 51 | 55
score on a scale
  Week 52 | 0.3 (1.73) | 0.2 (1.61) | -0.4 (1.74) | -0.3 (1.31)
  Week 78: number analyzed (Participants) | 53 | 52 | 50 | 55
  Week 78 | -0.5 (2.58) | -0.1 (1.54) | -0.4 (1.69) | -0.9 (1.92)
  Week 104: number analyzed (Participants) | 38 | 38 | 39 | 41
  Week 104 | -1.4 (3.29) | -0.9 (2.77) | -1.1 (2.56) | -1.3 (2.35)
  >=Week 117: number analyzed (Participants) | 2 | 1 | 4 | 1
  >=Week 117 | -3.0 (4.24) | 0.0 (NA) — SD does not apply when n = 1. | 0.3 (2.06) | 0.0 (NA) — SD does not apply when n = 1.

7. Secondary Outcome: Change in Muscles of the Thigh
Description: Magnetic resonance imaging (MRI) was planned to be used to characterize changes in muscles of the thigh in a subset of patients.
Time Frame: up to 1 year, up to 2 years
Population: No participants were analyzed. The optional MRI assessment was not initiated as the study was stopped.
Arm/Group | BYM338/Bimagrumab 10 mg/kg | BYM338/Bimagrumab 3 mg/kg | BYM338/Bimagrumab 1 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Patients With Anti-BYM338 Antibodies
Description: Investigated the development of immunogenicity against BYM338.
Time Frame: end of double-blind treatment (up to 8 months)
Population: Safety set: The safety set consisted of all participants who were assigned to treatment in the core study and who received at least one dose of study drug during the extension. Only those participants who provided a sample were analyzed.
Measure: Number; unit: Participants
Arm/Group | BYM338/Bimagrumab 10 mg/kg | BYM338/Bimagrumab 3 mg/kg | BYM338/Bimagrumab 1 mg/kg | Placebo
Number analyzed (Participants) | 38 | 40 | 38 | 39
Participants | 0 | 1 | 0 | 2

ADVERSE EVENTS:
Time Frame: Adverse events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All adverse events reported in this record are from date of First Patient First Treatment until Last Patient Last Visit, up to 14 months.
Groups:
- Pooled Active Treatment Groups: Participants from all 3 BYM338 groups
Arm/Group | BYM338/Bimagrumab 10 mg/kg | BYM338/Bimagrumab 3 mg/kg | BYM338/Bimagrumab 1 mg/kg | Placebo | Pooled Active Treatment Groups
All-Cause Mortality (participants affected / at risk) | 1/53 | 1/52 | 1/51 | 2/55 | 3/156
Serious Adverse Events (participants affected / at risk) | 12/53 | 10/52 | 7/51 | 8/55 | 29/156
Other Adverse Events (participants affected / at risk) | 40/53 | 46/52 | 38/51 | 43/55 | 124/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BYM338/Bimagrumab 10 mg/kg (N=53) | BYM338/Bimagrumab 3 mg/kg (N=52) | BYM338/Bimagrumab 1 mg/kg (N=51) | Placebo (N=55) | Pooled Active Treatment Groups (N=156)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Oesophageal achalasia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 1 | 1 | 3
Sepsis (Infections and infestations) | 1 | 0 | 0 | 2 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 2
Avulsion fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Inclusion body myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 2 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 2
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Peripheral venous disease (Vascular disorders) | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BYM338/Bimagrumab 10 mg/kg (N=53) | BYM338/Bimagrumab 3 mg/kg (N=52) | BYM338/Bimagrumab 1 mg/kg (N=51) | Placebo (N=55) | Pooled Active Treatment Groups (N=156)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 4 | 0 | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 9 | 5 | 9 | 5 | 23
Seasonal allergy (Immune system disorders) | 0 | 0 | 3 | 1 | 3
Nasopharyngitis (Infections and infestations) | 0 | 4 | 1 | 0 | 5
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 4 | 4 | 10
Contusion (Injury, poisoning and procedural complications) | 9 | 7 | 12 | 8 | 28
Fall (Injury, poisoning and procedural complications) | 30 | 36 | 30 | 34 | 96
Foot fracture (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 4 | 4
Injury (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 1 | 4
Joint injury (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0 | 3
Laceration (Injury, poisoning and procedural complications) | 1 | 7 | 4 | 6 | 12
Ligament sprain (Injury, poisoning and procedural complications) | 5 | 2 | 2 | 3 | 9
Limb injury (Injury, poisoning and procedural complications) | 3 | 1 | 1 | 0 | 5
Skin abrasion (Injury, poisoning and procedural complications) | 6 | 7 | 4 | 5 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 6 | 6 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 3 | 1 | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 8 | 3 | 1 | 15
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 3 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 1 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4 | 2 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 2 | 0 | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 5 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 5 | 3 | 2 | 9
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 3 | 1
Headache (Nervous system disorders) | 1 | 2 | 4 | 3 | 7
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 3 | 2
Acne (Skin and subcutaneous tissue disorders) | 2 | 1 | 3 | 1 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0 | 2 | 3 | 5
Rash (Skin and subcutaneous tissue disorders) | 2 | 3 | 3 | 1 | 8
Haematoma (Vascular disorders) | 2 | 0 | 2 | 4 | 4
Hypertension (Vascular disorders) | 5 | 2 | 2 | 1 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.